CLINICAL TRIAL: NCT02570477
Title: Fecal Microbiota Transplantation (FMT) for Moderate to Severe Clostridium Difficile Infection (CDI): A Randomised Study With Concurrent Stool Microbiota Assessment (FMT-CDI-RCT Study)
Brief Title: FMT for Moderate to Severe CDI: A Randomised Study With Concurrent Stool Microbiota Assessment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMT-CDI-RCT
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fecal Microbiota Transplantatio (Active Comparator): Fecal Microbiota Transplantation of stool from healthy donor to recipient.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Standard Therapy (Active Comparator): 125mg Vancomycin four times per day
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation — Healthy donor is screened and donates feces. It will then be diluted with sterile saline, blended and filtered. Supernatant will be infused to recipient.
  Other Names: FMT infusion
  Arms: Fecal Microbiota Transplantatio
Drug: Vancomycin — 125mg Vancomycin four times per day
  Arms: Standard Therapy

SUMMARY:
Clostridium difficile infection (CDI) is a leading cause of hospital-associated gastrointestinal illness, associated with significant morbidity and mortality and has a high burden on health-care system. The incidence of CDI has increased to epidemic proportion worldwide over the past decade. Community-acquired CDI, elderly and hospitalized patients receiving antibiotics are the main group at risk for developing CDI.

Currently, the first-line treatment for C. difficile-associated diarrhea includes cessation of the antibiotic implicated in the development of CDI, treatment with metronidazole or vancomycin and recently Fidaxomicin which is yet to be available in Hong Kong. However, disease recurrence is an increasing problem and 20% to 60% of patients experience at least one recurrence within a few weeks of completion of antibiotic treatment. Moreover, an increasing number of patients who require life-saving emergency colectomy experience persistent CDI after surgery. Until recently, an effective treatment against recurrent CDI is not available. Generally, repeated and extended courses of vancomycin are prescribed.

Fecal microbiota transplantation (FMT) defined as infusion of feces from healthy donors to affected subjects has attracted great interest in recent years and is now recommended as the most effective therapy for CDI not responding to standard therapies. Systematic reviews of prospective trials, case series and one randomized controlled trial have shown an overall cure rate of close to 100%. More than 50% of patients stated they would have FMT as their preferred first treatment option if CDI were to recur.

This proposal aims to investigate the efficacy of FMT as first line therapy in patients with severe CDI and to assess changes in the fecal microbiota after FMT using pyrosequencing techniques.

DETAILED DESCRIPTION:
Clostridium difficile infection (CDI) is a leading cause of hospital-associated gastrointestinal illness, associated with significant morbidity and mortality and has a high burden on health-care system. The incidence of CDI has increased to epidemic proportion worldwide over the past decade. Community-acquired CDI, elderly and hospitalized patients receiving antibiotics are the main group at risk for developing CDI 1.

Currently, the first-line treatment for C. difficile-associated diarrhea includes cessation of the antibiotic implicated in the development of CDI, treatment with metronidazole or vancomycin and recently Fidaxomicin which is yet to be available in Hong Kong2. However, disease recurrence is an increasing problem and 20% to 60% of patients experience at least one recurrence within a few weeks of completion of antibiotic treatment. Moreover, an increasing number of patients who require life-saving emergency colectomy experience persistent CDI after surgery. Until recently, an effective treatment against recurrent CDI is not available. Generally, repeated and extended courses of vancomycin are prescribed3.

Fecal microbiota transplantation (FMT) defined as infusion of feces from healthy donors to affected subjects has attracted great interest in recent years and is now recommended as the most effective therapy for CDI not responding to standard therapies 4. Systematic reviews of prospective trials, case series and one randomized controlled trial have shown an overall cure rate of close to 100% 5, 6. More than 50% of patients stated they would have FMT as their preferred first treatment option if CDI were to recur 7.

While FMT has been proven to be effective in refractory CDI, the role of FMT as first-line therapy in a subset of patients with severe CDI, or high risk features for severe CDI has not been studied. These are generally patients in whom the risk of colectomy and mortality is exceedingly high. In addition, the mechanism of FMT in CDI is not completely clear, and limited data are available on the effects of FMT on the microbiota post FMT. It has been suggested that CDI results in deficiencies in fecal flora composition, particularly of Bacteroides and Firmicutes, and these deficiencies in the microbiota facilitate colonization with C. difficile. Microarray analysis in small number of subjects has shown a major shift in the patients' microbiota after donor-feces infusion toward that of the donors8. The experimental tools required for in depth analysis of the intestinal microbiota are now becoming available. This study aims to investigate the efficacy of FMT as first line therapy in patients with moderate to severe CDI and to assess changes in the fecal microbiota after FMT using pyrosequencing techniques.

ELIGIBILITY:
Inclusion Criteria:

1. C. difficile infection defined as diarrhea (≥3 soft, loose or watery stools per day for at least 2 consecutive days or ≥8 soft or loose stools in 48 hours) and a positive stool test for C. difficile toxin; and
2. Age ≥ 18; and
3. Written informed consent obtained

Exclusion Criteria:

1. The presence of human immunodeficiency virus (HIV) infection with a CD4 count of less than 240
2. Pregnancy
3. GI Bleeding
4. Acute coronary syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants cured without relapse within 10 weeks after the initiation of therapy | 10 weeks
  Relapse is defined as diarrhea with a positive stool test for C. difficile toxin. An adjudication committee members who are not aware of the study-group assignment will make final decision on which patients are considered cured.

SECONDARY OUTCOMES:
30-day mortality rate | 30 days
  mortality rate is measured.
30-day colectomy rates | 30 days
  Colectomy rates is measured.
Number of day of hospital stay | up to 30 days
  The total hospital day is measured.
Changes in the stool microbiota after FMT measured using pyrosequencing | 30 days
  We will do pyrosequencing using the study stool samples from patients and donors

CONTACTS AND LOCATIONS:
Overall Officials: Siew Chien Ng, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zuo T, Wong SH, Lam K, Lui R, Cheung K, Tang W, Ching JYL, Chan PKS, Chan MCW, Wu JCY, Chan FKL, Yu J, Sung JJY, Ng SC. Bacteriophage transfer during faecal microbiota transplantation in Clostridium difficile infection is associated with treatment outcome. Gut. 2018 Apr;67(4):634-643. doi: 10.1136/gutjnl-2017-313952. Epub 2017 May 24. PMID 28539351